CLINICAL TRIAL: NCT02329795
Title: Image-derived Prediction of Response to Chemo-radiation in Patients With Glioblastoma
Brief Title: Image-derived Prediction of Response to Chemo-radiation in Glioblastoma
Acronym: IDEPREG
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Lundemann Jensen, Ph.d.-fellow, M.Sc., Rigshospitalet, Denmark
Other Study IDs: 192/13
Record Dates: First submitted 2014-12-16; First posted 2015-01-01 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Standard chemoradiotherapy: Group to receive 60 Gy radiotherapy in 30 fractions with concomitant and adjuvant temozolomide.
  Interventions: Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: Radiotherapy — 60 Gy in 30 fractions, 5 days a week, modulated arc therapy.
Drug: Temozolomide — Concomitant: 75 mg/m2 5 days a week from start of radiotherapy. Adjuvant: 150/200 mg/m2 in 5 days per 28 days in 6 months.
  Other Names: Temodar

SUMMARY:
This study seeks to investigate if advanced image-analysis of diagnostic scans, can be used to predict how aggressive brain tumors (glioblastoma) respond to standard chemo- and radiation treatment.

DETAILED DESCRIPTION:
Generally, response prediction models seeks to predict time to an event, e.g. time-to-progression and/or overall survival. The aim of this study is to explore the feasibility of establishing an individualized response model, that, based on several morphologic, physiologic and metabolic parameters extracted from computed tomography (CT), positron emission tomography (PET) and magnetic resonance imaging (MRI), is able to predict the tumor response at the level of an imaging voxel, using machine learning techniques.

Imaging modalities include MRI, PET/CT with 18F-fluroethyltyrosine (18F-FET), and PET/MRI with 64Cu-diacetyl-bis(N4-methylthiosemicarbazone) (64Cu-ATSM).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, primary supratentorial glioblastoma (WHO grade IV).

Exclusion Criteria:

* No informed consent can be obtained
* Inability to undergo MRI examination, due to metal implants, pacemaker etc.
* Not eligible for Stupp-regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary glioblastoma, eligible for chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of predicted response | 3 months post radiotherapy
  Tumor response is measured as contrast-enhancing tumor on T1-weighted MRI and by metabolic active tumor using 18F-fluroethyl-tyrosine (FET)-PET. Pre-treatment risk map is constructed using machine learning methods and compared to post-treatment scans.

SECONDARY OUTCOMES:
DICE-similarity coefficient and percentage overlap of 64Cu-ATSM and contrast-enhanced T1-weighted MRI | 3 months post radiotherapy
  Pre-chemoradiotherapy 64Cu-ATSM-PET is used as a surrogate marker for hypoxia and compared to treatment response, measured as contrast-enhancing tumor on T1-weighted MRI
Correlation (volume and maximum values) between lactate and hypoxia | 1 week before start of chemoradiotherapy
  Lactate measured by MR spectroscopy is compared to metabolic uptake of 64Cu-ATSM-PET

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Section for Radiotherapy, Rigshospitalet, Copenhagen, Denmark